CLINICAL TRIAL: NCT01576497
Title: Optimal Number of To-and-fro Motion in EUS-guided Fine Needle Aspiration for Pancreatic Masses in Terms of Suction or Without Suction: Prospective Randomized Single Blinded Trial
Brief Title: Optimal Number of To-and-fro Motion in EUS-guided Fine Needle Aspiration for Pancreatic Masses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Do Hyun Park, Assistant Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2012-0018
Record Dates: First submitted 2012-04-07; First posted 2012-04-12 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2012-04

CONDITIONS: Pancreatic Masses
Keywords: EUS, EUS-FNA, Pancreatic masses
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Suction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-FNA with suction (Active Comparator): EUS-FNA with suction/10, 15, 20 to-and-fro motion vs. EUS-FNA with suction/10, 15, 20 to-and-fro motion Visual assessment as stoping rule: 20 to-and-fro motion at different site will be performed when EUS-FNA sampling with 10, 15, 20 to-and-fro motion is unsatisfactory.
  Interventions: Device: EUS-FNA with suction
- EUS-FNA without suction (Active Comparator): EUS-FNA with suction/10, 15, 20 to-and-fro motion vs. EUS-FNA without suction/10, 15, 20 to-and-fro motion Visual assessment as stoping rule: 20 to-and-fro motion at different site will be performed when EUS-FNA sampling with 10, 15, 20 to-and-fro motion is unsatisfactory.
  Interventions: Procedure: EUS-FNA; Device: EUS-FNA without suction

INTERVENTIONS:
Procedure: EUS-FNA — EUS-FNA with suction/10, 15, 20 to-and-fro motion vs. EUS-FNA without suction/10, 15, 20 to-and-fro motion Visual assessment as stoping rule: 20 to-and-fro motion at different site will be performed when EUS-FNA sampling with 10, 15, 20 to-and-fro motion is unsatisfactory.
  Other Names: FNA with or without suction
  Arms: EUS-FNA without suction
Device: EUS-FNA with suction — For this prospective single-blinded randomized trial, two 10cc syringes was prepared. Two syringe was provided as same performance. However, one syringe is falsely made as suction syringe (fake one). During EUS-FNA, two syringe is randomly assigned and loaded by a nurse. Thus, operator was blinded which syringe is with suction or without suction.
  Other Names: FNA with suction
  Arms: EUS-FNA with suction
Device: EUS-FNA without suction — For this prospective single-blinded randomized trial, two 10cc syringes was prepared. Two syringe was provided as same performance. However, one syringe is falsely made as suction syringe (fake one). During EUS-FNA, two syringe is randomly assigned and loaded by a nurse. Thus, operator was blinded which syringe is with suction or without suction.
  Other Names: FNA without suction
  Arms: EUS-FNA without suction

SUMMARY:
EUS-FNA is the standard of care for diagnosing pancreatic masses. According to the operator's preference, EUS-FNA with suction or without suction technique has been used. To date, little is known about optimal number of to-and-fro motion during each needle pass. As usual 10-15 to-and-fro motions was used for EUS-FNA with suction technique. Theoretically, more number of to-and-fro motions may be required in EUS-FNA without suction. In this circumstance, the contamination of blood in specimen and possible adverse event may occur. To determine optimal number of to-and-fro motion in EUS-guided FNA for pancreatic masses in terms of with suction or without suction, this prospective single-blinded randomized trial was conducted.

DETAILED DESCRIPTION:
For this prospective single-blinded randomized trial, two 10cc syringes was prepared. Two syringe was provided as same performance. However, one syringe is falsely made as suction syringe (fake one). During EUS-FNA, two syringe is randomly assigned and loaded by a nurse. Thus, operator was blinded which syringe is with suction or without suction.

First hypothesis: There is difference in the diagnostic accuracy of pancreatic masses according to EUS-FNA with suction or without suction/ different number of to-and-fro motion.

Second hypothesis: There is difference in the amount of blood in samples obtained by EUS-FNA with suction or without suction/ different number of to-and-fro motion.

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years Solid pancreatic mass lesions

Exclusion Criteria:

* Age < 19 years Coagulopathy Unable to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 year
  The diagnostic accuracy of pancreatic masses at each sample according to EUS-FNA with suction or without suction/ different number of to-and-fro motion will be measured.
  Diagnostic accuracy of EUS-FNA with suction and 10, 15, and 20 to-and-fro motion vs.Diagnostic accuracy of EUS-FNA without suction and 10, 15, and 20 to-and-fro motion.

SECONDARY OUTCOMES:
Blood contamination in each sample | 1 year
  The amount of blood contamination at each sample according to EUS-FNA with suction or without suction/ different number of to-and-fro motion will be measured.
  The amount of blood contamination of EUS-FNA with suction and 10, 15, and 20 to-and-fro motion vs. The amount of blood contamination of EUS-FNA without suction and 10, 15, and 20 to-and-fro motion.

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea